CLINICAL TRIAL: NCT06052332
Title: Efficacy and Safety of Conventional Neoadjuvant Therapy Versus Total Neoadjuvant Therapy in Older Patients With Locally Advanced Rectal Cancer: a Multicentre, Open-label, Randomised Pragmatic Clinical Trial
Brief Title: Efficacy and Safety of Conventional Neoadjuvant Therapy Versus Total Neoadjuvant Therapy in Older Patients With Locally Advanced Rectal Cancer
Acronym: SHAPERS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IJB-SHAPERS-ODN-013
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Rectal Cancer; Older People
Keywords: rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional arm (Experimental): * SCRT (5 fractions of 5 Gy)
  * Surgery (according to the principle of TME) or watch & wait
  * Optional adjuvant chemotherapy
  OR
  * LCCRT (25-28 fractions of 1.8-2.0 Gy each +/- a boost to the primary tumour and involved lymph nodes, for a total of 50-56 Gy of radiation combined with either continuous infusion fluorouracil or capecitabine) followed by
  * Surgery (according to the principles of TME) or watch & wait, followed by
  * Optional adjuvant chemotherapy
  Interventions: Radiation: Short course radiotherapy; Drug: Adjuvant chemotherapy (optional); Procedure: Total mesorectal excision; Radiation: Long course chemoradiotherapy
- TNT arm (Active Comparator): Rapido regimen:
  * SCRT (5 fractions of 5 Gy)
  * Up to 18 weeks of oxaliplatin based chemotherapy (mFOLFOX6 or CAPOX)
  * Surgery (according to the principle of TME) or "watch & wait"
  Or
  Rapido light regimen:
  * SCRT
  * Up to 12 weeks of oxaliplatin based chemotherapy
  * Surgery or "watch & wait"
  Or
  OPRA with induction chemotherapy (INCT-CRT) regimen:
  * Up to 16 weeks of oxaliplatin-based chemotherapy
  * CRT (25-28 fractions of 1.8-2.0 Gy each +/- a boost to the primary tumour and involved lymph nodes, for a total of 50-56 Gy of radiation combined with either continuous infusion ﬂuorouracil or capecitabine)
  * Surgery or "watch & wait"
  Or
  OPRA with consolidation chemotherapy (CRT-CNCT) regimen:
  * CRT
  * Up to 16 weeks of oxaliplatin-based chemotherapy
  * Surgery or "watch & wait"
  Interventions: Procedure: Total mesorectal excision; Combination Product: Total neoadjuvant therapy

INTERVENTIONS:
Radiation: Short course radiotherapy — Patients will receive 5 daily fractions of radiotherapy. Each fraction will consist of 5 Gy for a total dose of 25 Gy.
  Arms: Conventional arm
Drug: Adjuvant chemotherapy (optional) — The choice of the adjuvant chemotherapy is to the investigator's discretion.
  Arms: Conventional arm
Procedure: Total mesorectal excision — Surgery must be performed according to the principles of total mesorectal excision. A "watch & wait" approach is allowed for those subjects who have clinical complete response according to the local assessment.
Combination Product: Total neoadjuvant therapy — The choice of the TNT is left to the investigator's discretion.
  If RAPIDO:
  * SCRT (5 fractions of 5 Gy), followed by
  * Up to 18 weeks of oxaliplatin based chemotherapy (mFOLFOX6 or CAPOX)
  If RAPIDO light:
  * SCRT (5 fractions of 5 Gy), followed by
  * Up to 12 weeks of oxaliplatin based chemotherapy (mFOLFOX6 or CAPOX)
  If OPRA with induction chemotherapy:
  * Up to 16 weeks of oxaliplatin-based chemotherapy (mFOLFOX6 or CAPOX), followed by
  * CRT (25-28 fractions of 1.8-2.0 Gy each +/- a boost to the primary tumour and involved lymph nodes, for a total of 50-56 Gy of radiation combined with either continuous infusion ﬂuorouracil or capecitabine)
  If OPRA with consolidation chemotherapy:
  * CRT (25-28 fractions of 1.8-2.0 Gy each +/- a boost to the primary tumour and involved lymph nodes, for a total of 50-56 Gy of radiation combined with either continuous infusion ﬂuorouracil or capecitabine) followed by
  * Up to 16 weeks of oxaliplatin-based chemotherapy (mFOLFOX6 or CAPOX)
  Arms: TNT arm
Radiation: Long course chemoradiotherapy — Patients will receive 25-28 fractions of 1.8-2.0 Gy each +/- a boost to the primary tumour and involved lymph nodes, for a total of 50-56 Gy of radiation combined with either continuous infusion fluorouracil or capecitabine
  Arms: Conventional arm

SUMMARY:
The SHAPERS study is a multicentre, open-label, randomised, pragmatic clinical trial, comparing standard-of-care neoadjuvant treatment options for older (i.e., ≥70 years) subjects with high-risk stage II and stage III rectal cancer.

DETAILED DESCRIPTION:
The SHAPERS study is a multicentre, open-label, randomised, pragmatic clinical trial, comparing standard-of-care neoadjuvant treatment options for older (i.e., ≥70 years) subjects with high-risk stage II and stage III rectal cancer.

Subjects meeting all eligibility criteria will be randomised in a 1:1 ratio to either the conventional arm or the TNT arm (The study design is shown in figure 3.1 and 3.2).

Conventional arm consists of:

* SCRT (5 fractions of 5 Gy), followed by
* Surgery (according to the principles of TME) or watch & wait, followed by
* Optional adjuvant chemotherapy OR
* LCCRT (25-28 fractions of 1.8-2.0 Gy each +/- a boost to the primary tumour and involved lymph nodes, for a total of 50-56 Gy of radiation combined with either continuous infusion fluorouracil or capecitabine) followed by
* Surgery (according to the principles of TME) or watch & wait, followed by
* Optional adjuvant chemotherapy

TNT arm Different treatment regimens can be used in the TNT arm including Rapido, Rapido light, OPRA INCT-CRT or OPRA CRT-CNCT. The regimen to use will be decided by the investigator and will need to be declared before randomisation. No switch between regimens is allowed during the study treatment period.

The Rapido regimen consists of:

* SCRT (5 fractions of 5 Gy), followed by
* Up to 18 weeks of oxaliplatin based chemotherapy (mFOLFOX6 or CAPOX), followed by
* Surgery (according to the principle of TME) or "watch & wait".

The Rapido light regimen consists of:

* SCRT (5 fractions of 5 Gy), followed by
* Up to 12 weeks of oxaliplatin based chemotherapy (mFOLFOX6 or CAPOX), followed by
* Surgery (according to the principle of TME) or "watch & wait".

The OPRA with induction chemotherapy (INCT-CRT) regimen, consists of:

* Up to 16 weeks of oxaliplatin-based chemotherapy (mFOLFOX6 or CAPOX), followed by
* CRT (25-28 fractions of 1.8-2.0 Gy each +/- a boost to the primary tumour and involved lymph nodes, for a total of 50-56 Gy of radiation combined with either continuous infusion ﬂuorouracil or capecitabine) followed by
* Surgery (according to the principle of TME) or "watch & wait"

The OPRA with consolidation chemotherapy (CRT-CNCT) regimen consists of:

* CRT (25-28 fractions of 1.8-2.0 Gy each +/- a boost to the primary tumour and involved lymph nodes, for a total of 50-56 Gy of radiation combined with either continuous infusion ﬂuorouracil or capecitabine) followed by
* Up to 16 weeks of oxaliplatin-based chemotherapy (mFOLFOX6 or CAPOX), followed by
* Surgery (according to the principle of TME) or "watch & wait".

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 70 years old
2. ECOG performance status (PS):

   * ≤1 if age > 75 years old
   * ≤2 if age ≤ 75 years old
3. Histologically or cytologically confirmed adenocarcinoma of the rectum
4. Distal border of the tumour below the peritoneal reflection and within 15 cm of the anal verge
5. Operable stage III or high-risk stage II rectal cancer (high-risk tumours defined as those having ≥1 of the following features: T4, mesorectal fascia (MRF) involvement/threatening [i.e.,tumour within 1 mm of the MRF], extramural venous invasion). Patient with involvement of lateral pelvic lymph nodes are also eligible.
6. Adequate bone marrow function as defined below:

   * Absolute neutrophil count ≥1,500/µL
   * Haemoglobin ≥9 g/dL
   * Platelets ≥100,000/µL
7. Adequate liver function as defined below:

   * Serum total bilirubin ≤1.5 x ULN. In case of known Gilbert's syndrome <3xUNL is allowed
   * AST (SGOT) and ALT (SGPT) ≤2.5 x ULN
   * Alkaline phosphatase ≤2.5 x ULN
8. Adequate renal function as defined by estimated glomerular filtration rate (GFR) ≥30 mL/min/1.73m² (according to the CKD-EPI 2021 equation).
9. Absence of clinical conditions that in the opinion of the investigator, would contraindicate neoadjuvant therapy and/or surgery.
10. Signed Informed Consent form (ICF) obtained prior to any study related procedure.
11. Male subjects with partners of childbearing potential must agree to use condom during the course of this study and for at least 6 months after the last administration of study drugs.

Exclusion Criteria:

1. Extensive growth into cranial part of the sacrum (above S2/3 junction) or the lumbosacral nerve roots indicating that surgery will never be possible even if substantial tumour down-sizing is achieved.
2. Presence of metastatic disease or recurrent rectal tumour.
3. Presence of grade ≥2 peripheral neuropathy according to the Common Toxicity Criteria for Adverse Events (CTCAE) v.5.0.
4. Significant medical, neuro-psychiatric, or surgical condition, currently uncontrolled by treatment, which, in the principal investigator's opinion, may interfere with completion of the study.
5. Any contraindication to pelvic irradiation as evaluated by the investigator.
6. Known hypersensitivity reactions to the study drugs or to any excipients, premedications or non-investigational medicinal products or concomitant medications.
7. Any investigational anti-cancer therapy other than the protocol specified therapies (participation in other prospective studies which do not imply any specific intervention may be allowed after discussion with the Study Chair).
8. Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment.
9. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke, myocardial infarction, unstable angina, congestive heart failure (grade III or IV as classified by the New York Heart Association), or serious cardiac arrhythmia requiring medication within the past 6 months.
10. Complete dihydropyrimidine dehydrogenase (DPD) deficiency.
11. Any previous treatment for rectal cancer.
12. Use of brivudine, sorivudine or their chemically related analogues.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | At 3 years after randomisation
  Overall survival (OS) will be calculated from randomisation to death from any cause.
Progression-free survival | At 3 years after randomisation
  Progression-free survival (PFS) will be calculated from randomisation to any of the following events: unresectable tumour due to local tumour progression, R2 resection of the primary tumour, loco-regional recurrence after an R0/R1 resection, distant metastases, or death from any cause.
Any grade peripheral sensory neuropathy | At 3 years after randomisation
  Any grade peripheral sensory neuropathy as assessed by the investigator according to the NCI-CTCAE v5.0 will be analysed.
Grade ≥3 toxicities during treatment | At 3 years after randomisation
  Grade ≥3 toxicities during treatment (i.e., from the 1st day of treatment until the EOT visit) as assessed by the investigator according to the NCI-CTCAE v5.0 will be analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Sclafani, Study Chair — Jules Bordet Institute
Locations (19):
- Belgium (19):
  - ZAS Antwerpen, Antwerp, Antwerpen
  - UZA Antwerpen, Edegem, Antwerpen
  - AZ Turnhout, Turnhout, Antwerpen
  - Institut Jules Bordet, Anderlecht, Brussels Capital
  - Chirec Delta, Auderghem, Brussels Capital
  - CHU Saint-Pierre, Brussels, Brussels Capital
  - CHU Brugmann, Brussels, Brussels Capital
  - UZ Gent, Ghent, East Flanders
  - AZ Nikolaas, Sint-Niklaas, East Flanders
  - Hôpital de Jolimont, Haine-Saint-Paul, Hainaut
  - Epicura, Hornu, Hainaut
  - CHU Ambroise Pare, Mons, Hainaut
  - CHU de Liège - Sart Tilman, Liège, Liège
  - CHA Libramont, Libramont, Luxemburg
  - Grand Hôpital De Charleroi, Charleroi, Namur
  - CHU Charleroi, Charleroi, Namur
  - CHU UCL Namur, Godinne, Namur
  - CHR Sambre et Meuse (site Meuse), Namur, Namur
  - CHU St Elisabeth, Namur, Namur

REFERENCES:
- [Derived] Saude-Conde R, Vandamme T, De Backer M, Martinive P, Covas A, Deleporte A, Dermine A, Forget F, Geboes K, Gilliaux Q, Gokburun Y, Gonne E, Joye I, Lecomte S, Liberale G, Lybaert W, Moretti L, Mortier L, Mupingu Mwanawa S, Puleo F, Saad ED, Sinapi I, Annemans L, Buyse M, Sclafani F. Efficacy and safety of short-course radiotherapy versus total neoadjuvant therapy in older rectal cancer patients: a randomised pragmatic trial (SHAPERS). ESMO Gastrointest Oncol. 2024 Jun 5;4:100067. doi: 10.1016/j.esmogo.2024.100067. eCollection 2024 Jun. PMID 41648032